CLINICAL TRIAL: NCT00070642
Title: ProMune™ (CPG 7909 Injection) With or Without Chemotherapy for the Treatment of Stage III b/c or IV Melanoma: A Randomized, Multi-Center, Open Label, Parallel Group, Active-Controlled, Phase II/III Study
Brief Title: CPG 7909 Injection in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C023; CO23, A8501023
Record Dates: First submitted 2003-10-06; First posted 2003-10-08 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Melanoma
Keywords: Immunotherapy, skin cancer
MeSH Terms: conditions — Carcinoma; Melanoma; Skin Neoplasms | interventions — ProMune; Dacarbazine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CPG 7909 Injection plus chemotherapy (Experimental): CPG 7909 Injection plus DTIC
  Interventions: Drug: CPG 7909 Injection; Drug: dacarbazine
- Chemotherapy alone (Active Comparator): dacarbazine
  Interventions: Drug: Chemotherapy
- CPG 7909 Injection 10 mg (Experimental)
  Interventions: Drug: CPG 7909 Injection
- CPG 7909 Injection 40 mg (Experimental)
  Interventions: Drug: CPG 7909 Injection

INTERVENTIONS:
Drug: CPG 7909 Injection — CPG 7909 Injection administered subcutaneously at a dose of 40 mg weekly.
  Other Names: ProMune, PF-3512676
  Arms: CPG 7909 Injection plus chemotherapy
Drug: dacarbazine — dacarbazine 850mg/m2 in three-week cycles until disease progression
  Other Names: DTIC
  Arms: CPG 7909 Injection plus chemotherapy
Drug: Chemotherapy — Chemotherapy in three-week cycles until disease progression:
  dacarbazine 850mg/m2
  Other Names: DTIC
  Arms: Chemotherapy alone
Drug: CPG 7909 Injection — CPG 7909 Injection administered subcutaneously at a dose of 10 mg weekly.
  Other Names: ProMune, PF-03512676
  Arms: CPG 7909 Injection 10 mg
Drug: CPG 7909 Injection — CPG 7909 Injection administered subcutaneously at a dose of 40 mg weekly.
  Other Names: ProMune, PF-03512676
  Arms: CPG 7909 Injection 40 mg

SUMMARY:
To determine the safety, tolerability and effects of CPG 7909 (the study drug) when given with chemotherapy to patients with melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma that is metastatic.
* Measurable disease according to the RECIST criteria.
* Karnofsky Performance Status of > 70.

Exclusion Criteria:

* Prior treatment with anti-neoplastic biologic or chemotherapy for recurrent or metastatic disease (except one course of adjuvant immunotherapy and/or adjuvant chemotherapy other than DTIC).
* Suspected or known CNS metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Phase II: Assess the anti-neoplastic activity, as determined by overall response rate (complete plus partial responses) according to the RECIST criteria. | indeterminate
Phase III: Evaluate and compare the survival time of the two treatment groups, as selected in Phase II. | Indeterminate

SECONDARY OUTCOMES:
Phase III: Assess the overall response rate | indeterminate
Asses the degree of clinical benefit defined as the proportion of patients experiencing complete and partial responses as well as stable disease. | indeterminate
Determine the duration of response. | indeterminate
Determine the time to progression | indeterminate
Assess the pharmacokinetic profile and immunopharmacodynamic response to CPG 7909 Injection alone or in combination with DTIC, or DTIC alone (immunopharmacodynamic response only). | indeterminate
Describe the tolerability of CPG 7909 Injection alone, CPG 7909 Injection in combination with DTIC vs. DTIC alone | indeterminate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CO23&StudyName=CPG%207909%20Injection%20in%20Melanoma